CLINICAL TRIAL: NCT04364074
Title: Acute Impact of Probiotic Supplementation on Endothelial Function in Adults
Brief Title: Acute Probiotic Supplementation and Endothelial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Michael E. Widlansky, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 37096
Record Dates: First submitted 2020-04-24; First posted 2020-04-27 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Coronary Artery Disease; Hypertension; Hyperlipidemias; Peripheral Vascular Diseases; Cerebral Arterial Diseases
MeSH Terms: conditions — Coronary Artery Disease; Hypertension; Hyperlipidemias; Peripheral Vascular Diseases; Cerebral Arterial Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GoodBelly Probiotic (Experimental): Subjects randomized to this arm consume one serving of the Goodbelly lactobacillus plantarum 299v probiotic
  Interventions: Dietary Supplement: Goodbelly
- Placebo (Placebo Comparator): Subjects randomized to this arm consume one serving of the Goodbelly that does not contain lactobacillus plantarum 299v
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Goodbelly — Consumption of 1 serving of Goodbelly probiotic daily for 6 weeks. This will be followed by an observation period for 6 weeks during which the subjects will not consume Goodbelly.
  Other Names: Goodbelly probiotic
  Arms: GoodBelly Probiotic
Dietary Supplement: Placebo — To prepare the placebo, the dietitian will first heat a water bath to 80 degrees Celsius. This removes the lactobacillus plantarum 299v from the probiotic drink
  Other Names: Goodbelly Probitoic
  Arms: Placebo

SUMMARY:
One in every two deaths in the United States is caused by cardiovascular disease. Despite strong mechanistic links established between a diet rich in lipids and the pathogenesis of cardiovascular disease, therapeutic advances have focused on reduction in either ingestion or synthesis of cholesterol, and reduction in dietary trans and saturated fatty acids and triglycerides. Even in the setting of aggressive high potency statin therapy and global cardiovascular risk reduction efforts, most clinical trials reveal a significant residual cardiovascular risk with, at best, only 30% reduction in major adverse cardiovascular events. There exists a significant unmet clinical need for identifying novel therapies for the prevention and treatment of cardiovascular disease. This requires identification of additional contributory processes to cardiovascular disease pathogenesis, so that mechanism-based interventions may be developed. Endothelial dysfunction is a pathological state in which there is systemic inflammation of vascular endothelium with consequent expression of pro-vasoconstrictive mediators, thrombotic and atherogenic tendencies. Endothelial dysfunction precedes the development of atherosclerosis and portends an increased risk of future adverse cardiovascular events. Endothelial dysfunction, therefore, can serve as a "barometer" of future cardiovascular risk. Measurement of Flow-mediated dilation ( FMD) is widely accepted as a method to assess vascular endothelial function.

DETAILED DESCRIPTION:
Researchers at MCW have discovered a new pathway that links the type of bacteria present in the intestines to the severity of heart attacks. This discovery of a relationship between intestinal bacteria, bacterial metabolites, and severity of heart attacks means that for the first time, we may be able to determine a person's probability of having a heart attack via non-conventional risk factors. This may provide opportunities for novel diagnostic tests as well as a potential for therapeutic intervention. The link between gut microbiota and the severity of heart attacks may also lead to novel therapeutic approaches (probiotics, non-absorbable antibiotics) to prevent heart attacks from happening. Our pilot study has demonstrated that supplementation of Lactobacillus plantarum 299v (Lp299v) for 6 weeks to adults with a history of coronary artery disease showed improvement in endothelial function. Whether acute ingestion of a single drink containing Lp299v supplementation favorably impacts vascular endothelial function is not known. The study proposed will test the hypothesis that supplementation of Lp299v favorably impacts vascular endothelial function after ingestion of a single supplement containing Lp299v.

Specific Aim 1 will determine the acute impact of probiotic supplementation on endothelial cell function as measured by brachial artery flow mediated dilation (FMD)

Specific Aim 2 will determine the impact of acute probiotic supplementation on blood biomarkers for inflammation.

Specific Aim 3 will be to determine the impact of baseline constitution of intestinal microbiota (assessed by stool microbiome) on change in FMD as a result of acute response to probiotic supplementation.

Specific Aim 4 will be to determine the impact of baseline constitution of intestinal microbiota (assessed by stool microbiome) on change in levels of blood markers for inflammation as a result of acute response probiotic supplementation.

ELIGIBILITY:
Inclusion Criteria:

Have at least one of the following conditions:

* Hypertension
* Hyperlipidemia
* Diabetes mellitus (Type 1 or Type 2)
* Peripheral vascular disease
* Cerebrovascular disease
* Cardiovascular disease.

Exclusion Criteria:

* Unstable angina or myocardial infarction by history, ECG, and/or enzymatic criteria within 1 month of enrollment.
* LV dysfunction as defined by an LV ejection fraction documented as < 45% within 1 year of enrollment by an echocardiogram, MRI, or nuclear imaging.

Uncontrolled hypertension with blood pressure greater than 170/100 mmHg at the screening visit.

* Known history of chronic renal insufficiency, liver dysfunction, or cancer besides non-melanoma skin carcinomas or localized prostate cancer requiring systemic treatment within five years of enrollment.
* Known history of cognitive impairment or inability to follow study procedures
* Patient with an implanted defibrillator or permanent pacemaker on which the potential participant is known to rely upon for greater than 50% of ventricular depolarizations.
* Patients who received probiotics, prebiotics, and antibiotics in the last 12 weeks.
* Patients with dosing changes of vasoactive medications and HMG-CoA reductase inhibitors in the 6 weeks prior to enrollment.
* Pregnancy
* Patients who are currently taking Vitamin K antagonists such as coumadin, warfarin.
* Those who are daily drinkers.
* Patients with gastrointestinal diseases that might alter the impact of a probiotic (e.g. status post colectomy, short gut syndrome, or inflammatory bowel disease)

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
change in baseline flow mediated dilation (FMD) after probiotic consumption | from baseline to 24 hours after consumption and approximately 7 days after consumption
  This is a measurement of endothelial function in the brachial artery

SECONDARY OUTCOMES:
Interleukin-6 | from baseline to 24 hours after consumption and approximately 7 days after consumption
  Circulating marker of inflammation
Interleukin-8 | from baseline to 24 hours after consumption and approximately 7 days after consumption
  Circulating marker of inflammation
Interleukin-12 | from baseline to 24 hours after consumption and approximately 7 days after consumption
  Circulating marker of inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Wauwatosa, Wisconsin, United States